CLINICAL TRIAL: NCT01909427
Title: A Randomized, Placebo-controlled Double-blind, Multicenter, Phase 2 Dose Ranging Study To Assess The Efficacy And Safety of CNTO 6785 In Subjects With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: An Efficacy And Safety Study of CNTO 6785 In Participants With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100935; CNTO6785ARA2001 (Other: Janssen Research & Development, LLC); 2012-003629-40 (EudraCT Number)
Record Dates: First submitted 2013-07-10; First posted 2013-07-26 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Active rheumatoid arthritis despite methotrexate therapy; CNTO 6785; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo/CNTO 6785 200 mg+Methotrexate (MTX) (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: CNTO 6785 200 mg; Drug: Methotrexate (MTX)
- CNTO 6785 200 mg+MTX (Experimental)
  Interventions: Drug: CNTO 6785 200 mg; Drug: Methotrexate (MTX)
- CNTO 6785 100 mg+MTX (Experimental)
  Interventions: Drug: CNTO 6785 100 mg; Drug: Methotrexate (MTX)
- CNTO 6785 50 mg+MTX (Experimental)
  Interventions: Drug: CNTO 6785 50 mg; Drug: Methotrexate (MTX)
- CNTO 6785 15 mg+MTX (Experimental)
  Interventions: Drug: CNTO 6785 15 mg; Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Placebo — Placebo subcutaneous injections (SC) every 4 weeks through Week 12
  Arms: Placebo/CNTO 6785 200 mg+Methotrexate (MTX)
Drug: CNTO 6785 200 mg — CNTO 6785 200 mg SC every 4 weeks from Week 16 through Week 28
  Arms: Placebo/CNTO 6785 200 mg+Methotrexate (MTX)
Drug: CNTO 6785 200 mg — CNTO 6785 200 mg SC every 4 weeks through Week 28
  Arms: CNTO 6785 200 mg+MTX
Drug: CNTO 6785 100 mg — CNTO 6785 100 mg SC every 4 weeks through Week 28
  Arms: CNTO 6785 100 mg+MTX
Drug: CNTO 6785 50 mg — CNTO 6785 50 mg SC every 4 weeks through Week 28
  Arms: CNTO 6785 50 mg+MTX
Drug: CNTO 6785 15 mg — CNTO 6785 15 mg SC every 4 weeks through Week 28
  Arms: CNTO 6785 15 mg+MTX
Drug: Methotrexate (MTX) — MTX at the same stable dose through Week 32, that participants were receiving prior to screening.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of CNTO6785 in participants with active rheumatoid arthritis (RA) despite methotrexate (MTX) therapy.

DETAILED DESCRIPTION:
This is a randomized (participants are assigned to treatment by chance), double-blind (participants and study personnel will not know which treatments are being given), placebo-controlled (a placebo appears identical to a study drug but has no active ingredients), multicenter study. The study will consist of 3 phases: a screening phase, a treatment phase, and a follow-up phase. Approximately 250 participants with active RA despite MTX therapy will be randomly assigned to receive placebo or CNTO 6785 during the double-blind treatment phase. The maximum period of active treatment will be 28 weeks. The maximum duration of study participation will be 44 weeks. Participant safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of rheumatoid arthritis (RA) (according to the revised 1987 criteria of the American Rheumatism Association) and have had RA for at least 6 months prior to the date of signing the informed consent at screening
* Have active RA defined study as persistent disease activity with both of the following criteria: at least 6 swollen and 6 tender joints using a 66/68 joint count at the time of screening and at baseline; and serum C-reactive protein (CRP) ≥ 0.8 mg/dL at screening or erythrocyte sedimentation rate (ESR) ≥ 28 mm in the first hour at screening or baseline
* Have been treated with and tolerated methotrexate (MTX) treatment at dosages from 7.5 to 25 mg/week, inclusive, for a minimum of 6 months prior to screening and must have a stable MTX dose for a minimum of 6 weeks prior to the first dosing with study agent

Exclusion Criteria:

* Has inflammatory diseases other than RA, that might confound the evaluation of the benefit of study agent therapy
* Has a diagnosis of fibromyalgia
* Has a recent history (within 12 months prior to screening) of uncontrolled, chronic disease including, but not limited to, pulmonary, psychiatric, and metabolic disturbances, cardiovascular, endocrine, neurological, hepatic, gastrointestinal, renal, hematological, or urological diseases that the investigator believes are clinically significant
* At screening, the results of laboratory tests must meet protocol-specified criteria
* Has ever received any approved or investigational biologic agent for a rheumatic indication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who achieve an ACR 20 response at Week 16 | Week 16
  American College of Rheumatology (ACR) 20 response is a >=20% improvement in rheumatoid arthritis (RA) symptoms.

SECONDARY OUTCOMES:
Change from baseline in DAS28 (CRP) at Week 16 | Baseline to Week 16
  DAS28 (using CRP [C-reactive protein]) is a measure of tender and swollen joints and the patient's assessment of disease activity.
The proportion of participants who achieve ACR 50 response at Week 16 | Week 16
  American College of Rheumatology (ACR) 50 response is a >=50% improvement in rheumatoid arthritis (RA) symptoms.
The proportion of participants who achieve ACR 20 response through Week 32 | Week 32
The proportion of participants who achieve ACR 50 response through Week 32 | Week 32
The proportion of participants who achieve ACR 70 response through Week 32 | Week 32
  American College of Rheumatology (ACR) 70 response is a >=70% improvement in rheumatoid arthritis (RA) symptoms.
Change from baseline of DAS28 (CRP) through Week 32 | Baseline to Week 32
The proportion of participants with DAS28 (CRP) response through Week 32 | Week 32
  DAS28 (using CRP [C-reactive protein]) response is improvement from baseline, with >1.2 indicating a good or moderate response and <=0.6 indicating no response.
The proportion of participants with DAS28 (CRP) remission at Week 16 | Week 16
  DAS28 (using CRP [C-reactive protein]) remission is defined as a value of <2.6 on the Disease Activity Index, a measure of tender and swollen joints and the patient's assessment of disease activity.
The proportion of participants with DAS28 (CRP) remission at Week 32 | Week 32
Change from baseline in DAS28 (ESR) at Week 16 | Baseline to Week 16
  DAS28 (using erythrocyte sedimentation rate) is a measure of tender and swollen joints and the patient's assessment of disease activity.
Change from baseline in DAS28 (ESR) at Week 32 | Baseline to Week 32
Change from baseline in HAQ-DI score through Week 32 | Baseline to Week 32
  The Health Assessment Questionnaire-Disability Index (HAQ-DI) assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas, each scored from 0 (no difficulty) to 3 (inability to perform a task).
Change from baseline in SF-36 at Week 16 | Baseline to Week 16
  The SF-36 is a medical outcome study health measure and consists of 8 multi-item scales that are scored from 0 to 100, with higher scores indicating better health.
Change from baseline in SF-36 at Week 32 | Baseline to Week 32
Change from baseline in CDAI at Week 16 | Baseline to Week 16
  Clinical Disease Activity Index (CDAI) score is a derived score combining tender joints (28 joints), swollen joints (28 joints), Patient's Global Assessment of Disease Activity, and Physician's Global Assessments of Disease Activity.
Change from baseline in CDAI at Week 32 | Baseline to Week 32
Change from baseline in SDAI at Week 16 | Baseline to Week 16
  The Simplified Disease Activity Index (SDAI) score is a derived score combining tender joints (28 joints), swollen joints (28 joints), Patient's Global Assessment of Disease Activity, Physician's Global Assessments of Disease Activity, and CRP.
Change from baseline in SDAI at Week 32 | Baseline to Week 32
The proportion of participants with SDAI-based ACR/EULAR remission at Week 16 | Week 16
  The Simplified Disease Activity Index (SDAI)-based ACR/EULAR (European League Against Rheumatism) remission is defined as a SDAI value of <=3.3 at a visit.
The proportion of participants with SDAI-based ACR/EULAR remission at Week 32 | Week 32
The proportion of participants with Boolean-based ACR/EULAR remission at Week 16 | Week 16
  Boolean-based ACR/EULAR remission is achieved if all of the following 4 criteria at that visit are met: tender joint count (68 joints) <=1; swollen joint count (66 joints) <=1; CRP <=1 mg/dL; and Patient's Global Assessment of Disease Activity on VAS <=1 on a 0 to 10 scale.
The proportion of participants with Boolean-based ACR/EULAR remission at Week 32 | Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- Argentina (5):
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Córdoba
  - La Capital
  - San Juan
- Colombia (3):
  - Barranquilla
  - Bogotá
  - Medellín
- Czechia (2):
  - Jihlava
  - Prague
- Philippines (4):
  - Cebu
  - Iloilo City
  - Lipa City
  - Quezon City
- Poland (7):
  - Bydgoszcz
  - Grodzisk Mazowiecki
  - Lodz
  - Lublin
  - Poznan
  - Warsaw
  - Wroclaw
- Russia (9):
  - Barnaul
  - Kemerovo
  - Kursk
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Saint Petersburg
  - Yaroslavl
  - Yekaterinburg
- Thailand (2):
  - Bangkok
  - Chiang Mai